CLINICAL TRIAL: NCT01438021
Title: Characterization of the Pharmacokinetics and Efficacy of Intraventricular Methotrexate Continuously Delivered Via a Mini Pump for Treatment of Leptomeningeal Disease
Brief Title: Continuous Intraventricular Methotrexate in Treating Patients With Leptomeningeal Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09201; NCI-2011-03006 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-09-19; First posted 2011-09-21 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Leptomeningeal Metastases
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — Methotrexate; merphos

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (intraventricular chemotherapy) (Experimental): Patients receive intraventricular methotrexate continuously on days 1-14. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: pharmacological study; Drug: methotrexate

INTERVENTIONS:
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Drug: methotrexate — Given intraventricularly
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX

SUMMARY:
This pilot clinical trial studies continuous intraventricular methotrexate in treating patients with leptomeningeal disease. Drugs used in chemotherapy, such as methotrexate, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving drugs directly into the ventricles may be an effective treatment for patients with leptomeningeal disease

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the pharmacokinetics and efficacy of continuous intraventricular methotrexate infusion in the treatment of leptomeningeal disease.

SECONDARY OBJECTIVES:

I. Describe the dose limiting toxicities. II. Describe the pharmacodynamics of continuously delivered intraventricular methotrexate.

III. Assess for response.

OUTLINE:

Patients receive intraventricular methotrexate continuously on days 1-14. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with leptomeningeal carcinomatosis (from solid tumors)
* Subjects with lymphomatous or leukemic meningitis
* The effects of methotrexate on the developing fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following the conclusion of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she will be excluded from the study and should inform her treating physical immediately
* Karnofsky Performance Status greater than 70%
* All subjects must have the ability to understand and the willingness to sign a written informed consent
* We will exclude subjects who have had prior intrathecal/intraventricular therapy with methotrexate within 6 months

Exclusion Criteria:

* Prior therapy with methotrexate for management of leptomeningeal disease
* Subjects with evidence of hydrocephalous
* Subjects with intraparenchymal lesions or bulky disease
* Subjects with ventriculoperitoneal shunt in place
* Previous history of whole brain radiation therapy
* Subjects who, in the opinion of the principal investigator, may not be able to comply with the safety monitoring requirements of the study will not be included in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy of continuously delivered intraventricular methotrexate | Day 3 after start of treatment
  The concentration of methotrexate in the brain parenchyma will be determined with microdialysis probe placed next to the ventricle.
Pharmacokinetics of continuous intraventricular infusion of methotrexate | Day 14 after start of treatment
  Determined by measuring brain interstitial levels of methotrexate using microdialysis catheters, lumbar cerebral spinal fluid (CSF) levels (a distant site) of methotrexate via a lumbar drain during the inpatients phase, ventricular CSF levels of methotrexate using the Ommaya reservoir, and systemic levels of methotrexate in the blood.

SECONDARY OUTCOMES:
Response rate of continuous intraventricular methotrexate infusion | Day 42 after start of treatment
Toxicities of continuous intraventricular methotrexate infusion | Day 3 after start of treatment
Pharmacodynamics of continuously delivered intraventricular methotrexate | Day 42 after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mike Chen, MD, Principal Investigator — City of Hope Medical Center